CLINICAL TRIAL: NCT01113463
Title: A Phase 2 Open-Label Study of the Efficacy of TPI 287 in Patients With Glioblastoma Multiforme That Has Recurred or Progressed Following Prior Therapy With Radiation Plus Temozolomide
Brief Title: TPI 287 in Patients With Recurrent Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0759; NCI-2011-01303 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-27; First posted 2010-04-30 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Brain Cancer
Keywords: Brain Tumor; Central Nervous System; CNS; Glioblastoma Multiforme; GBM; TPI 287; Radiation Therapy; Temozolomide; Chemotherapy; taxanes
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPI 287 (Experimental): TPI 287 Starting dose 160 mg/m^2 intravenous (IV) every 3 weeks
  Interventions: Drug: TPI 287

INTERVENTIONS:
Drug: TPI 287 — Starting dose of 160 mg/m^2 as a 60-minute (± 10 minutes) IV infusion once every 3 weeks, (i.e., 1 cycle = 21 days).

SUMMARY:
The goal of this clinical research study is to learn if TPI 287 can help to control glioblastoma. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

TPI 287 is designed to block a protein that causes cancer cells to resist the effects of chemotherapy. By blocking the protein, the drug may be able to cause the cancer cells to shrink or stop growing.

Bevacizumab will be given to patients that are found to have brain damage, as described below. It is designed to block the growth of new blood vessels. It may help to lower the amount of brain damage related to tumor tissue death and help limit the symptoms of this condition.

Study Drug Administration:

On Day 1 of each 21-day study "cycle," you will receive TPI 287 by vein over about 1 hour.

If you experience intolerable side effects, the dose of TPI 287 may be lowered. Your doctor will tell you more about lowering a dose due to side effects.

To help prevent an allergic reaction to TPI 287, you will also receive the following drugs:

* Benadryl® (diphenhydramine) by vein over 30 minutes, 30-60 minutes before you receive TPI 287
* Cimetidine by vein over 30 minutes, 30-60 minutes before you receive TPI 287
* Either dexamethasone or methylprednisolone (taken by mouth 12 and 6 hours before you receive TPI 287; or by vein over 30 minutes at about 30-60 minutes before you receive TPI 287)

If you have an MRI scan that shows evidence of brain damage related to the tumor tissue death after you have received TPI 287 for two infusions, you will be eligible to receive bevacizumab. On Day 1 of Cycle 3 and beyond, if you are eligible, you will receive bevacizumab by vein over about 60-90 minutes.

Study Visits:

At each study visit, you will be asked about any drugs you may be taking and about any side effects you may have experienced.

On Day 1 of Cycle 1:

* Your weight and vital signs will be measured.
* If your doctor thinks it is needed, blood (about 1 tablespoon) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests

On Day 15 of every even-numbered cycle (Cycles 2, 4, 6, and so on), you will have an MRI scan to check the status of the disease.

Length of Study:

You will be on study for up to 6 months. You may continue to receive the study drug for as long as you are benefiting. You will be taken off study if the disease gets worse or if you experience intolerable side effects.

If you are eligible and you receive it, you may continue to receive bevacizumab for as long as you are benefiting. You will be taken off bevacizumab if the disease gets worse or if you experience intolerable side effects.

End-of-Treatment Visit:

Within 28 days after you stop receiving the study drug, you will have an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have an MRI scan to check the status of the disease if you did not have one within 6 weeks before the end-of-treatment visit.

Long-Term Follow-Up:

Every 3 months for up to 1 year after you stop receiving the study drug, you will be called and asked about how you are feeling. Each phone call will last about 5-10 minutes.

This is an investigational study. TPI 287 is not FDA approved or commercially available. It is currently being used for research purposes only. Bevacizumab is FDA approved and commercially available for the treatment of brain tumors. The use of bevacizumab for brain damage related to the tumor tissue death is investigational.

Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histological or cytological documentation of GBM. Patients will be eligible if the original histology was lower grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made.
2. Patients must have supratentorial GBM that has radiographic recurrence or progression following prior radiation therapy and temozolomide for GBM or lower grade glioma, or the appearance of new lesions on scan, or clinical or neurologic worsening despite stable disease on the last 2 scans.
3. Patients must have measurable disease on radiologic scan.
4. Patients must be >/= 18 years of age.
5. Patients must have a Karnofsky performance status >/= 60%.
6. Patients must have adequate bone marrow as evidenced by an absolute neutrophil count >/=1,500/uL and a platelet count >/=100,000/uL.
7. Patients must have adequate renal function as evidenced by serum creatinine <= the upper limit of normal (ULN)
8. Patients must have adequate hepatic function as evidenced by serum total bilirubin </= 2.0 mg/dL and aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) </= 3 times the ULN.
9. Patients must have recovered from the effects of any prior surgery, radiotherapy or other chemotherapy with any therapy related adverse events revolved to </= grade 1, and at least 12 weeks must have elapsed from the completion of radiotherapy, and 3 weeks from the last dose of Temozolomide.
10. Women of child-bearing potential (includes women who are menopausal for less than 1 year and not surgically sterilized) must have a negative urine or serum pregnancy test at screening.
11. Sexually active patients must agree to use adequate contraception (two barrier methods) for the duration of the study.
12. Patients or their legal representative must be able to read, understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Patients who have received more than one course of radiation therapy or more than a total dose of 65 grey (Gy). Patients may have received radiosurgery as part of the initial therapy (i.e., in addition to one course of radiation therapy); however, the dose used for the radiosurgery counts against the total dose limit listed above.
2. Patients who have had a second surgery for recurrent disease who have no radiologically apparent residual disease (contrast-enhanced MRI imaging must have been performed within 24-48 hours post-operatively).
3. Patient who have received any cytotoxic chemotherapy for treatment of GBM other than temozolomide (Gliadel trademarked as part of the initial therapy is permitted). However, patients who have received prior biologic therapy will be eligible.
4. Patients who are receiving concurrent enzyme-inducing anti-epileptic drugs (EIAEDs) (e.g., carbamazepine, oxcarbazepine, phenytoin, fosphenytoin, phenobarbital and primidone) or who received EIAEDs within 2 weeks prior to the first dose of study drug.
5. Patients who are not on a stable or decreasing steroid dose for the previous week prior to the study enrollment.
6. Patients with an active infection or with a fever >/= 38.5°C within 3 days prior to the study enrollment.
7. Patients who have history of prior malignancy within the past 5 years except for curatively treated non-melanoma skin cancer or cervical intra-epithelial neoplasia for which the patient has been disease-free for at least 3 years.
8. Patients with Grade 2 or higher peripheral neuropathy.
9. Patients with New York Heart Association(NYHA) Class 3 or 4 congestive heart failure.
10. Patients with known HIV or Hepatitis B or C.
11. Patients who are pregnant or lactating.
12. Patients with any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the patient's ability to sign the ICF or his/her ability to cooperate and participate in the study, or to interfere with the interpretation of the results.
13. Patients who have received prior bevacizumab therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Conrad, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 27, 2010 to August 09, 2011. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: The study stopped enrollment of participants since a competing study with the drug combination was planned.
Period: Overall Study
Arm/Group | TPI 287
Started | 17
Completed | 12
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: Insufficient enrollment to perform any meaningful statistical analysis, therefore study terminated early.
Arm/Group | TPI 287
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 61 [31 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 6 Months
Description: PFS defined as number of participants alive without documented evidence of disease progression ("progression free") at 6 months. Progression-free survival calculated from the date of Day 1 Cycle 1 to the date that criteria for progression of disease is first seen. Progression is defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months (following nine 21-day cycles)
Population: Intent to treat population included all eligible subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 17
participants | 0

2. Secondary Outcome: Number of Participants by Response Criteria
Description: Complete Response (CR): Complete disappearance all measurable & evaluable disease. No new lesions or evidence of non-evaluable disease. Partial Response (PR): >/= 50% decrease under baseline in sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease, nor new lesions. Stable/No Response: Does not qualify for CR, PR, or progression. The designation of Stable/No Response requires a minimum of 12 weeks duration. Progression: 25% increase in sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). Unknown: Progression not been documented & one or more measurable or evaluable sites have not been assessed.
Time Frame: Response obtained between days 15 and 21 of every even cycle and/or when clinically indicated, up to 6 months (approximately 9 completed cycles)
Population: Intent to treat population included all eligible subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 17
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable/No Response | 6
  Progression | 10
  Unknown | 1

ADVERSE EVENTS:
Time Frame: Adverse event reporting from Day 1, cycle 1 to 30 days after last dose of treatment drug. Study period was May 26, 2010 to June 30, 2011.
Arm/Group | TPI 287
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 17/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TPI 287 (N=17)
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 1
Allergic Rhinitis (Immune system disorders) | 1
Change in SGPT/SGOT (Metabolism and nutrition disorders) | 4 — aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT)
Ataxia (Nervous system disorders) | 2
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increase (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 8
Gait/Walking Difficulty (Musculoskeletal and connective tissue disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hemoglobin Changes (Blood and lymphatic system disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with Normal Anc (Lung - Pneumonia) (Infections and infestations) | 1
Infection with Normal ANC (Urinary Tract Nos) (Infections and infestations) | 2
Insomnia (General disorders) | 1
Leukocytes, low (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 3
Memory Impairment (Nervous system disorders) | 1
Altered Mental Status (Nervous system disorders) | 2 — Anxiety, Mood Alteration
Mucositis (Gastrointestinal disorders) | 1 — Mucositis (Clinical Exam) Oral Cavity
Muscle Weakness (Whole Body/Generalized) (Musculoskeletal and connective tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 — Neutrophils/granulocytes (ANC/AGC) low, Neutrophil Count Decreased
Pain (General disorders) | 5 — Pain, Extremity-Limb and other
Petechiae (Blood and lymphatic system disorders) | 1
Platelet Count Decreased (Blood and lymphatic system disorders) | 3
Psychosis (Nervous system disorders) | 1
Rigors/Chills (General disorders) | 1
Sensory Loss (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 1
Speech Impairment (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
Not enough subjects were enrolled to perform any meaningful statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No